CLINICAL TRIAL: NCT03271437
Title: Flash Open Trial With Therapists In Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Trauma Institute & Child Trauma Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-1003
Record Dates: First submitted 2017-08-31; First posted 2017-09-05 (Actual); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Trauma, Psychological
MeSH Terms: conditions — Psychological Trauma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PC-trained therapists (Experimental)
  Interventions: Behavioral: PC-based Flash
- EMDR-trained therapists (Experimental)
  Interventions: Behavioral: EMDR-based Flash

INTERVENTIONS:
Behavioral: PC-based Flash — Progressive counting with Flash technique
  Arms: PC-trained therapists
Behavioral: EMDR-based Flash — Eye movement desensitization and reprocessing with Flash technique
  Arms: EMDR-trained therapists

SUMMARY:
This study will test the eye movement desensitization and reprocessing (EMDR) based Flash technique and a progressive counting (PC) based variant. EMDR-trained therapists will be trained in the standard Flash, and PC-trained therapists will be trained in PC Flash. In each group they will try it with a minor upsetting memory, and then with two more significant upsetting memories. Participants will use the subjective units of distress scale (SUDS) to rate distress pre- and post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Therapist trained by Trauma Institute & Child Trauma Institute in EMDR or PC

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-09-15 (Estimated); Primary Completion 2017-11-30 (Estimated); Study Completion 2017-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in SUDS following treatment | Pre-treatment, immediately post-treatment, one week post-treatment, and one month post-treatment
  Subjective units of distress scale

CONTACTS AND LOCATIONS:
Overall Officials: Ricky Greenwald, PsyD, Principal Investigator — Trauma Institute & Child Trauma Institute
Locations (1):
- Trauma Institute & Child Trauma Institute, Northampton, Massachusetts, United States